CLINICAL TRIAL: NCT01276054
Title: Reducing the Incidence and Severity of Arm Lymphedema With Axillary Reverse Mapping and Implementation of a Lymphedema Screening and Intervention Program
Brief Title: Sentinel and/or Axillary Lymph Node Biopsy With or Without Axillary Reverse Mapping in Reducing Incidence and Severity of Arm Lymphedema in Stage 0-2 Patients.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: P.I. left
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1B-09-12; NCI-2010-02323 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-02

CONDITIONS: Lymphedema; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Technetium Tc 99m Sulfur Colloid; Methylene Blue; Indocyanine Green; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SNB plus ARM or ALND (+/- SNB) plus ARM (Experimental): Patients undergo sentinel lymph node biopsy (SNB) and/or axillary lymph node biopsy (ALND) using technetium Tc 99m sulfur colloid followed by methylene blue or indocyanine green solution tracer for localization of the arm lymph node. Patients then undergo an axillary reverse mapping.
  Interventions: Radiation: technetium Tc 99m sulfur colloid; Drug: methylene blue; Drug: indocyanine green solution; Procedure: sentinel lymph node biopsy; Procedure: axillary lymph node biopsy; Procedure: bioimpedance spectroscopy; Procedure: quality-of-life assessment; Other: lymphedema management
- SNB or ALND (+/- SNB) (Active Comparator): Patients undergo SNB and/or ALND using technetium Tc 99m sulfur colloid followed by methylene blue or indocyanine green solution tracer for localization of the arm lymph node.
  Interventions: Radiation: technetium Tc 99m sulfur colloid; Drug: methylene blue; Drug: indocyanine green solution; Procedure: sentinel lymph node biopsy; Procedure: axillary lymph node biopsy; Procedure: bioimpedance spectroscopy; Procedure: quality-of-life assessment

INTERVENTIONS:
Radiation: technetium Tc 99m sulfur colloid — Given intradermally and periareolarly
  Other Names: Tc 99m Sulfur Colloid; Tc-99m SC
Drug: methylene blue — Given subcutaneously
  Other Names: Azul de Metileno; Azul Metile; Blu di Metilene; MB
Drug: indocyanine green solution — Given subcutaneously
  Other Names: IC-GREEN; ICG solution
Procedure: sentinel lymph node biopsy — Undergo sentinel lymph node biopsy
  Other Names: sentinel node biopsy
Procedure: axillary lymph node biopsy — Undergo axillary lymph node biopsy
  Other Names: axillary node biopsy
Procedure: bioimpedance spectroscopy — Correlative studies
  Other Names: BIS
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: lymphedema management — Undergo axillary reverse mapping
  Arms: SNB plus ARM or ALND (+/- SNB) plus ARM

SUMMARY:
Lymph node biopsy followed by axillary reverse mapping may reduce the incidence and severity of arm lymphedema. This randomized phase II trial is studying how well sentinel and/or axillary lymph node biopsy with or without axillary reverse mapping works in reducing incidence and severity of lymphedema in patients with resectable stage 0-II breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To evaluate the ability of axillary reverse mapping (ARM) to reduce the incidence of lymphedema (LE) following axillary nodal staging. SECONDARY OBJECTIVES: I. To document the use of a standardized LE screening and LE level-specific management protocol on the outcome of LE among patients who develop LE. II. To document the relationship between limb volume measurements assessed by infrared laser perometry and bioelectrical impedance spectroscopy. OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients undergo sentinel lymph node biopsy (SNB) and/or axillary lymph node biopsy (ALND) using technetium Tc 99m sulfur colloid followed by methylene blue or indocyanine green solution tracer for localization of the arm lymph node. Patients then undergo and axillary reverse mapping. ARM II: Patients undergo SNB and/or ALND using technetium Tc 99m sulfur colloid followed by methylene blue or indocyanine green solution tracer for localization of the arm lymph node. After completion of study treatment, patients are followed up at 1-2 weeks, 3 months, and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0, I, and II Breast Cancer
* Not pregnant or breastfeeding
* Breast cancer or prophylactic mastectomy requiring axillary nodal staging
* Ability to read and/or comprehend consent form and questionnaires
* Ability to follow-up per protocol
* Unilateral axillary staging

Exclusion Criteria:

* Stage 3
* Previous axillary lymph node dissection
* Neoadjuvant chemotherapy or hormonal therapy exceeding greater than 30 days duration
* Allergy to blue dyes or iodine; NOTE: a non-blue dye or non-iodine-containing dye may be used in these patients
* Patients with implanted medical devices such as a pacemaker may undergo perometry, but not BIS (Bioelectrical Impedance Spectroscopy)
* Previous diagnosis of LE (lymphedema) of either extremity
* Bilateral axillary staging

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Holmes, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this trial opened in December 2010 and closed in June 2011 at which time the protocol was terminated due to the departure of the Principal Investigator.
Pre-assignment Details: The study has no pre-assignment.
Period: Overall Study
Arm/Group | SNB Plus ARM or ALND (+/- SNB) Plus ARM | SNB or ALND (+/- SNB)
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — No one to oversee trial after P.I. left | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SNB Plus ARM or ALND (+/- SNB) Plus ARM | SNB or ALND (+/- SNB) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Whether or Not a Patient Has Developed Grade 1+ LE
Description: LE is defined using the CTCAE v3 definition: a >5-10% increase in the inter-limb volume in the ipsilateral arm compared to the unaffected arm.
Time Frame: During the first year post-operatively
Population: Unable to analyze due to early termination of the study
Arm/Group | SNB Plus ARM or ALND (+/- SNB) Plus ARM | SNB or ALND (+/- SNB)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months from date on study
Arm/Group | SNB Plus ARM or ALND (+/- SNB) Plus ARM | SNB or ALND (+/- SNB)
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNB Plus ARM or ALND (+/- SNB) Plus ARM (N=2) | SNB or ALND (+/- SNB) (N=2)
Fatigue (General disorders) | 2 (3) | 2 (2)
Depression (Psychiatric disorders) | 1 (2) | 0 (0)
Edema - limbs (General disorders) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SNB Plus ARM or ALND (+/- SNB) Plus ARM (N=2) | SNB or ALND (+/- SNB) (N=2)
Pain (General disorders) | 2 (5) | 2 (4)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 2 (4)
Edema (General disorders) | 2 (2) | 0 (0) — Mastectomy site
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (5)
Depression (Psychiatric disorders) | 1 (1) | 2 (6)
Malaise (General disorders) | 2 (4) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Study terminated early due to P.I. moving to another institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No